CLINICAL TRIAL: NCT03149471
Title: The Role of Endothelial Function Test in Risk Stratification for Early and Late Complications After Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Shlomi Matetzky, Director , Cardiac Intensive Care Unit, Sheba Medical Center
Other Study IDs: ENOPAT_PE
Record Dates: First submitted 2017-03-20; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal endothelial function: patients diagnosed with PE and have normal endothelial function test- RHI score >=1.67
  Interventions: Diagnostic Test: Endothelial dysfunction test
- Endothelial dysfunction group: patients diagnosed with PE and have endothelial function- RHI<1.67
  Interventions: Diagnostic Test: Endothelial dysfunction test

INTERVENTIONS:
Diagnostic Test: Endothelial dysfunction test — The endothelial function test will be assessed after 48 hours post admission and 1 year post discharge using the non-invasive Endo-PAT2000 device. The device is intended for use as a diagnostic aid in the detection of coronary artery endothelial dysfunction (positive or negative) using a reactive hyperemia procedure. It is based on the use of Peripheral Arterial Tone (PAT) signal technology, during a clinically established procedure, which measure post-ischemic vascular responsiveness following upper arm blood flow occlusion.

SUMMARY:
The aim of this study is to investigate the association between endothelial dysfunction, measured by RHI as assessed by the peripheral arterial tonometry method, and PE complications defined as re-event of PE or DVT, systemic embolism or all-cause mortality

DETAILED DESCRIPTION:
200 Patients will be identified through routine daily scanning of imaging records (CT, Echocardiography) for patients diagnosed with PE. Presenting signs and symptoms as well as clinical and imaging findings during the initial presentation and hospitalization will be incorporated into a computerized pre-specified electronic CRF. During hospitalization, an endothelial function test will be performed 48 hours post admission. A trained technician will perform the test using the EndoPAT device in order to assess patient RHI, a score less than 1.67 will be considerate as endothelial dysfunction. Patients will then be followed for pre-specified clinical events of up to 1 year post discharge and especially the development of chronic thromboembolic pulmonary disease, post thrombotic syndrome and clinical events. RHI will be assessed during 1-year follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Patient is hospitalized with the diagnosis of acute PE
3. Clinically stable patients.
4. Clinical diagnosis of PE based on CT scan or nuclear imaging.
5. Willing and able to sign informed consent

Exclusion Criteria:

1. Previous myocardial infarction during the last 3 months.
2. Planned surgery or PCI.
3. Inability to perform endothelial function test.
4. Current participation in clinical trial.
5. Substrate or drug abuse or alcohol consumption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 Stable patients hospitalized in ICCU or Cardiology department with a diagnosis of acute PE according to CT scanning or nuclear imaging
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Post PE complications | 2 years
  The aim of this study is to investigate the association between endothelial dysfunction, measured by RHI as assessed by the peripheral arterial tonometry method, and PE complications defined as re-event of PE or DVT, systemic embolism or all-cause mortality

SECONDARY OUTCOMES:
Augmentation Index (AI) | 2 years
  To investigate the association between arterial stiffness as measured by Augmentation Index and post PE complications.
HRV | 2 years
  To investigate the association between Heart Rate Variability and post PE complications.
Biochemistry | 2 years
  To assess the association between troponin levels to post PE complications

IPD SHARING:
Plan to Share IPD: No
No IPD plan

REFERENCES:
- [Background] Heit JA. The epidemiology of venous thromboembolism in the community. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):370-2. doi: 10.1161/ATVBAHA.108.162545. No abstract available. PMID 18296591
- [Background] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Background] Goldhaber SZ. Venous thromboembolism: epidemiology and magnitude of the problem. Best Pract Res Clin Haematol. 2012 Sep;25(3):235-42. doi: 10.1016/j.beha.2012.06.007. Epub 2012 Aug 9. PMID 22959540
- [Background] Centers for Disease Control and Prevention (CDC). Venous thromboembolism in adult hospitalizations - United States, 2007-2009. MMWR Morb Mortal Wkly Rep. 2012 Jun 8;61(22):401-4. PMID 22672974
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, Lohse CM, O'Fallon WM, Melton LJ 3rd. The epidemiology of venous thromboembolism in the community. Thromb Haemost. 2001 Jul;86(1):452-63. PMID 11487036
- [Background] Becattini C, Cohen AT, Agnelli G, Howard L, Castejon B, Trujillo-Santos J, Monreal M, Perrier A, Yusen RD, Jimenez D. Risk Stratification of Patients With Acute Symptomatic Pulmonary Embolism Based on Presence or Absence of Lower Extremity DVT: Systematic Review and Meta-analysis. Chest. 2016 Jan;149(1):192-200. doi: 10.1378/chest.15-0808. Epub 2016 Jan 6. PMID 26204122
- [Background] Cohen AT, Dobromirski M, Gurwith MM. Managing pulmonary embolism from presentation to extended treatment. Thromb Res. 2014 Feb;133(2):139-48. doi: 10.1016/j.thromres.2013.09.040. Epub 2013 Oct 14. PMID 24182642
- [Background] Axtell AL, Gomari FA, Cooke JP. Assessing endothelial vasodilator function with the Endo-PAT 2000. J Vis Exp. 2010 Oct 15;(44):2167. doi: 10.3791/2167. PMID 20972417
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Bonetti PO, Lerman LO, Lerman A. Endothelial dysfunction: a marker of atherosclerotic risk. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):168-75. doi: 10.1161/01.atv.0000051384.43104.fc. PMID 12588755
- [Background] Cai H, Harrison DG. Endothelial dysfunction in cardiovascular diseases: the role of oxidant stress. Circ Res. 2000 Nov 10;87(10):840-4. doi: 10.1161/01.res.87.10.840. PMID 11073878
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159